CLINICAL TRIAL: NCT05377268
Title: The Use of Machine Learning Detection of Lipohypertrophy to Improve Glycemic Variability
Brief Title: The Use of Ultrasound Detection of Lipohypertrophy to Improve Glycemic Control
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kenneth Madden, Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: H22-01168
Record Dates: First submitted 2022-05-05; First posted 2022-05-17 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus; Lipohypertrophy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Patients will be randomized and data interpreters will be blinded to two, randomized, alternating 14-day protocols where the patients will be advised by the nurse educator verbally and by written instruction (recorded on a standardized grid as in our lab's previous work, see Appendix)11 to inject insulin in sites of subclinical lipohypertrophy (LH protocol) or normal subcutaneous tissue (Normal protocol). During each protocol, each subject will have glycemic variability measured.
Who Masked: Participant, Investigator
Masking Description: The subject and the investigators will be blinded to the order of the two crossover protocols
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LH Protocol (Experimental): Patients will be randomized and data interpreters will be blinded to two, randomized, alternating 14-day protocols where the patients will be advised by the nurse educator verbally and by written instruction to inject insulin in sites of subclinical lipohypertrophy.
  Interventions: Procedure: LH Protocol
- Normal Protocol (Active Comparator): Patients will be randomized and data interpreters will be blinded to two, randomized, alternating 14-day protocols where the patients will be advised by the nurse educator verbally and by written instruction to inject insulin in sites of normal subcutaneous tissue.
  Outcomes measured will consist of mean glucose, glucose standard deviation around the mean value, percentage of time with glucose below 3 mmol/liter, and percentage of time spent with glicose above 10 mmol/liter. The device will be calibrated and placed by a trained research nurse. There will be a member of the rsearch team available 24 hours per day to answer subject questions.
  Interventions: Procedure: LH Protocol

INTERVENTIONS:
Procedure: LH Protocol — Patients will be randomized and data interpreters will be blinded to two, randomized, alternating 14-day protocols where the patients will be advised by the nurse educator verbally to inject insulin in sites of subclinical lipohypertrophy
  Other Names: 40 patients identified with subclinical lipohypertrophy in Phase 1 will be recruited to a randomized crossover design examining glycemic variability by glucose monitor.

SUMMARY:
Lipohypertrophy is swelling of the fatty tissue located below the skin ("subcutaneous tissue") where many patients with diabetes inject their insulin. Lipohypertrophy can sometimes be felt as firm swelling, lumps or small bumps near insulin injection sites. Previous studies have shown that injecting insulin into areas of lipohypertrophy can affect how insulin is absorbed, and can increase insulin requirements in patients. New data suggest that lipohypertrophy can be detected using ultrasound technology. The ultrasonographic presence of changes to the subcutaneous tissue without swelling that can be felt ("subclinical lipohypertrophy") and the effect of injecting insulin into these sites is unknown.

100 people will participate in the Phase 1 of this study. In the second phase of the study, 40 patients identified with subclinical lipohypertrophy in Phase 1 will be asked to participate in the randomized study using crossover design by checking your glucose levels.

DETAILED DESCRIPTION:
Purpose:

In Phase 1: to use computer based technology to detect lipohypertrophy on portable ultrasound images.

In Phase 2: to demonstrate that injecting insulin into areas to be free of lipohypertrophy will have better glucose control as compared to injecting into areas demonstrated to have lipohypertrophy.

Eligibility:

You can participate in this study if:

* You have been diagnosed with Type 1 or Type 2 diabetes
* You are currently using injection of insulin daily or insulin pump for at least 2 years
* You are 19 years of age or older

You should not participate in this study if:

* You are taking a glucagon-like peptide medication
* You are currently using a systemic steroid agent (e.g. prednisone)
* You have history of a non-lipohypertrophic skin disease in the insulin injection area
* You are not fluent in English (unless accompanied by a translator)

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of Type 1 or Type 2 diabetes mellitus
* Current treatment with a minimum of one insulin injection daily or insulin pump for at least 2 years

Exclusion Criteria:

* Subjects taking a glucagon-like peptide-1 agonist or a systemic glucocorticoid
* Past history of a non-lipohypertrophic dermatological condition in the insulin injection site area

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of lipohypertrophy by US machine | First 12 months of the study
  Validation of machine algorithm, such as a web-based convolutional network to detect lipohypertrophy on portable ultrasound images.
  Each image will be evaluated by an experience ultrasonographer (Dr.Areshnikoff0 and labelled as either having the presence or absence of lipohypertrophy.

CONTACTS AND LOCATIONS:
Locations (1):
- Vancouver General Hospital Diabetes Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided